CLINICAL TRIAL: NCT04940273
Title: Intervention of Spontaneous Hyperventilation in Patients With Aneurysmal Subarachnoid Hemorrhage: the Feasibility of Drug Therapy and Its Impact on Cerebral Blood Flow
Brief Title: Drug Intervention of Spontaneous Hyperventilation in Patients With Aneurysmal Subarachnoid Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, department head, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2021-001
Record Dates: First submitted 2021-05-26; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Hyperventilation; Aneurysmal Subarachnoid Hemorrhage; Cerebral Blood Flow
Keywords: spontaneous hyperventilation; aneurysmal subarachnoid hemorrhage; cerebral blood flow; remifentanil; partial pressure of carbon dioxide
MeSH Terms: conditions — Hyperventilation; Subarachnoid Hemorrhage | interventions — Remifentanil; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- remifentanil (Experimental): Continuous infusion of remifentanil at a dose of 0.02、0.04、0.06、0.08 ug/kg/min for 30 minutes in sequence.
  Interventions: Drug: Remifentanil Injection [Ultiva]

INTERVENTIONS:
Drug: Remifentanil Injection [Ultiva] — Continuous infusion of remifentanil at a dose of 0.02、0.04、0.06、0.08 ug/kg/min for 30 minutes in sequence.
  Other Names: remifentanil hydrochloride for injection

SUMMARY:
Although spontaneous hyperventilation patients with aneurysmal subarachnoid hemorrhage closely associated with poor outcomes, the standard therapy remains unavailable. Remifentanil has the pharmacological characterization of respiratory inhibition, mainly prolonging the expiratory time and decreasing the respiratory rate while preserving the respiratory drive. The investigators hypothesis that spontaneous hyperventilation could be corrected by titrating the dose of remifentanil and cerebral blood flow will augment during this process.

DETAILED DESCRIPTION:
Evidence has shown a high incidence of spontaneous hyperventilation in patients with aneurysmal subarachnoid hemorrhage (aSAH), which is associated with poor outcomes. It's well established that the hypocapnia caused by hyperventilation leads to cerebral vasoconstriction, reduces the cerebral blood flow, and decreases the cerebral blood volume and intracranial pressure consequently. However, persistent cerebral vascular constriction increases the risk of cerebral ischemia; therefore, maintaining a partial pressure of arterial carbon dioxide (PaCO2) in the range of 35-40mmHg is recommended to minimize the hazard hypocapnia.

There's still no standard method to deal with spontaneous hyperventilation. Based on the pharmacology and clinical experience, remifentanil seems to be an ideal choice since it could inhibit the respiratory rate in a dose-dependent fashion. As one of the most used short-acting opioids, remifentanil could prolong the expiratory time, meanwhile not influencing the inspiratory time and respiratory drive, consequently decreasing respiratory rate and maintaining the tidal volume.

In this exploratory physiology study, the investigators will test the hypothesis that spontaneous hyperventilation could be suppressed by titrating the dose of remifentanil and could be realized as the target of PaCO2. The investigators will determine the optimal amount of remifentanil, which fulfills the criteria of efficacy and safety, and evaluate its effect on the cerebral blood flow velocity of both the middle cerebral artery and internal carotid artery.

ELIGIBILITY:
Inclusion Criteria:

* Aneurysmal subarachnoid hemorrhage, after craniotomy or clipping
* Arterial blood gas satisfy with PaCO2<35mmHg and pH>7.45
* Presence of an endotracheal tube
* Assisted ventilation mode,CPAP/PSV
* ICP monitoring

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Chronic obstructive pulmonary disease
* Allergy to opioids
* Clinically relevant hepatic or renal failure
* Hemodynamic instability
* TCD windows cannot detect cerebral blood flow
* Refuse to participate the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Explore the effective and safe dose of remifentanil to correct spontaneous hyperventilation in patients with aSAH | The PaCO2 (mmHg) at baseline and 30 minutes following each infusion rate adjustment (0.02、0.04、0.06、0.08μg/kg/min)
  The differences of partial pressure of carbon dioxide (PaCO2; mmHg) between the respective points (baseline and 30 minutes following each infusion rate adjustment of remifentanil) were recorded to determine the change of PaCO2 (mmHg).

SECONDARY OUTCOMES:
To explore the effect of remifentanil on the cerebral blood flow in patients with aSAH at the different dose | The MFV at baseline and 30 minutes following each infusion rate adjustment (0.02、0.04、0.06、0.08μg/kg/min)
  The differences of mean cerebral flow velocity (MFV) of middle cerebral artery and Internal carotid artery between baseline and 30 minutes following each infusion rate adjustment of remifentanil were recorded to determine the change of cerebral blood flow.

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Jian-Xin, MD, Study Director — Capital Medical University
Locations (1):
- ICU, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Su R, Zhou J, Zhu N, Chen X, Zhou JX, Li HL. Efficacy and safety of remifentanil dose titration to correct the spontaneous hyperventilation in aneurysmal subarachnoid haemorrhage: protocol and statistical analysis for a prospective physiological study. BMJ Open. 2022 Nov 9;12(11):e064064. doi: 10.1136/bmjopen-2022-064064. PMID 36351728